CLINICAL TRIAL: NCT01412892
Title: A Single Arm, Multicenter Phase II a Trial of RAD001 as Monotherapy in the Treatment of Neurofibromatosis 1 Related Internal Plexiform Neurofibromas That Cannot be Removed by Surgery
Brief Title: Use of RAD001 as Monotherapy in the Treatment of Neurofibromatosis 1 Related Internal Plexiform Neurofibromas
Acronym: NFitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P090502; 2010-023137-34 (EudraCT Number)
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Neurofibromatosis Type 1; Plexiform Neurofibroma; Neurofibromatoses
Keywords: Neurofibromatosis type 1; Everolimus; Plexiform neurofibromas; Rapamycin
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform; Neurofibromatoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): RAD001: Everolimus
  Interventions: Drug: RAD001: Everolimus

INTERVENTIONS:
Drug: RAD001: Everolimus — 10 mg of RAD001 will be self-administered orally once daily continuously for one year or until unacceptable toxicity or discontinuation from the study from any other reason.

SUMMARY:
Background:

Patients with the genetic disorder neurofibromatosis Type 1 (NF1) are at increased risk of developing tumors of the central and peripheral nervous system. These include plexiform neurofibromas. The conventional treatment of these internal plexiform neurofibromas is surgery. This surgery can be possible on a single and limited tumor. On the other hand these tumors are often surgically intractable due to their multiplicity and their infiltrating characteristics Increased activity of mammalian target of rapamycin(mTOR) protein is seen in neurofibromas. mTOR inhibitor rapamycin , or its derivatives such as everolimus may slow or stop tumor growth in patients with NF1.

Objectives:

Primary objectives To determine whether everolimus has an effect on the volume of surgically intractable and life-threatening internal plexiform neurofibromas in patients with neurofibromatosis 1.

Secondary objectives To determine whether everolimus has an effect on the number and the volume of cutaneous neurofibromas; to determine whether everolimus modify the signaling pathways in cutaneous neurofibromas.

Eligibility:

- Adults with neurofibromatosis type 1 with at least one internal plexiform neurofibroma, life-threatening or causing significant morbidity through compression of organs. This or these internal plexiform neurofibroma(s) should be intractable by surgery.

Design:

An open-label, single arm, non-randomized, single stage phase IIa study. Baseline phase: Baseline evaluations will be performed within 2 weeks, and up to a maximum of 4 weeks for specific exams, before the first dose of study drug.

Treatment phase/duration of treatment: All patients will be treated with RAD001 10 mg p.o daily dose for one year except in case of unacceptable toxicity, death, or discontinuation from the study for any other reason.

Follow-up phase: All patients will have two follow-up visits scheduled at 18 and 24 months after the first dose of the study drug to follow for adverse events (AEs) and serious adverse events (SAEs) that may have occurred after discontinuation from the study and for internal plexiform neurofibromas assessment.

Radiological review: All Magnetic Resonance Imaging (MRIs) obtained at baseline, during the treatment period and the follow-up period will be reviewed by the Neuroradiologist of the study.

DETAILED DESCRIPTION:
Neurofibromatosis 1 (NF1) is an autosomal dominant disease affecting 1 in 3000 to 1 in 4000 people. NF1 is characterized by multiple dermal neurofibromas, plexiform neurofibromas, malignant peripheral nerve sheath tumors (MPNST), and optic pathway gliomas, as well as by café-au-lait spots and abnormalities of the skeletal, cardiovascular and central nervous systems. The NF1 gene is located on chromosome 17q11.2, and its protein, neurofibromin, functions as a tumor suppressor.

People with NF1 have a decrease in life expectancy of 15 years, with MPNST as a leading cause of death in young adults. A specific phenotype at risk of mortality has been identified, patients with subcutaneous neurofibromas. Individuals with subcutaneous neurofibromas are more than 3 times as likely to have internal plexiform neurofibromas as others. Individuals with internal plexiform neurofibromas are 18 times more likely to develop MPNST than patients without internal plexiform neurofibromas. Beside MPNST, internal plexiform neurofibromas can be life-threatening or cause of significant morbidity through compression of organs mainly spine or nerve roots.

The conventional treatment of these internal plexiform neurofibromas is surgery. This surgery can be possible on a single and limited tumor. On the other hand these tumors are often surgically intractable due to their multiplicity and their infiltrating characteristics. In this context a medical treatment decreasing the size of these tumors would have its place with as short term aim to lower the consequence of compression and long-term aim to reduce the risk of malignant transformation.

NF1 is a consequence of the loss-of-function mutations in the NF1 tumor suppressor gene. The NF1-encoded protein, neurofibromin, functions as a Ras-GTPase activating protein (RasGAP). Accordingly, deregulation of Ras is thought to contribute to NF1 development. The mTOR pathway is tightly regulated by neurofibromin. mTOR is constitutively activated in both NF1-deficient primary cells and human tumors in the absence of growth factors. This aberrant activation depends on Ras and PI3 kinase, and is mediated by the phosphorylation and inactivation of the TSC2-encoded protein tuberin by AKT. Importantly, tumor cell lines derived from NF1 patients, and a genetically engineered cell system that requires Nf1-deficiency for transformation, are highly sensitive to the mTOR inhibitor rapamycin. Furthermore, the activation of endogenous Ras leads to constitutive mTOR signaling in this disease state, and in normal cells Ras is differentially required for mTOR signaling in response to various growth factors. Thus, the NF1 tumor suppressor is an indispensable regulator of TSC2 and mTOR. Ras plays a critical role in the activation of mTOR in both normal and tumorigenic settings.

mTOR inhibitor rapamycin potently suppresses the growth of aggressive NF1-associated malignancies in a genetically engineered murine model. In these tumors rapamycin does not function via mechanisms generally assumed to mediate tumor suppression, including inhibition of HIF-1 alpha and indirect suppression of AKT, but does suppress the mTOR target Cyclin D1. The mammalian target of rapamycin complex 1 inhibitor RAD001 (Everolimus) decreased growth 19% to 60% after 4 days of treatment in NF1 MPNST cell lines.

Finally, these data suggest that rapamycin, or its derivatives such as everolimus may represent a viable therapy for NF1. This proof of concept has been done in tuberous sclerosis where rapamycin was efficient to treat angiomyolipomas11.

The management of neurofibromatoses in France is coordinated by Pr. Pierre WOLKENSTEIN through the French National Referral Centre for Neurofibromatoses and a network, NF-France. The cohort followed up by the centre and its network is constituted of about 3000 patients and among them between 80 and 100 have life-threatening internal plexiform neurofibromas.

Therefore the investigators propose a trial to evaluate the efficacy of everolimus in surgically intractable and life-threatening internal neurofibromas in neurofibromatosis 1 based on the data of the literature and on our cohort.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NF1, according to NIH criteria, with internal plexiform neurofibroma (PN) and at least 1 of criteria for NF1:

  6 or more café-au-lait spots Freckling in the axilla or groin Optic glioma 2 or more Lisch nodules Distinctive bony lesion

  1-degree relative with NF1
* At least 1 inoperable PN(s) that has/have the potential to cause significant morbidity: Paravertebral lesions that could compromise the spinal cord Head and neck lesions that could compromise the airway or great vessels Brachial or lumbar plexus lesions that could cause nerve compression and loss of function Lesions that could result in major deformity (e.g., orbital lesions) or significant cosmetic problems Lesions of the extremity that cause limb hypertrophy or loss of function Painful lesions
* Complete resection of a PN with acceptable morbidity is not feasible OR patient refuses surgery OR the number of PNs leads to not feasible surgery according to the steering committee's site
* Measurable PN amenable to volumetric MRI analysis using fusion of images
* Measurable lesion (at least 3 cm in one dimension)
* Karnofsky >70%
* 18≤ Age ≤60
* absolute neutrophil count (ANC) ≥1.5x109/L, Platelets ≥100x109/L, Hb >9g/dL
* bilirubin: ≤1.5xULN, ALT and AST ≤2.5xULN unless evident Gilbert disease (amendment n°2). For patients with known liver metastases: AST and ALT ≤ 5xULN
* Creatinine ≤ 1.5xULN
* Life expectancy ≥ 2 years
* Cholesterol ≤300 mg/dL or ≤7.75 mmol/L and triglycerides ≤ 2.5x ULN
* Women of childbearing potential must have had a negative serum pregnancy test within 7 days and a negative urine pregnancy test within 72 hours prior to the administration of RAD001 start and must use an effective birth control method.
* Men should use condoms and their partner(s) use an effective birth control method
* A written informed consent obtained

Exclusion Criteria:

Patients who/with:

* have previously received mTOR inhibitors
* a known hypersensitivity to RAD001 or other rapamycin or to its excipients
* receiving chronic systemic treatment with corticosteroids or another immunosuppressive agent. (Dose equivalent to 10 mg/day of methylprednisone), topical steroids or organotherapy for bilateral adrenalectomy are acceptable
* a known history of HIV seropositivity
* acute viral hepatitis
* autoimmune hepatitis
* with an active, bleeding diathesis. Patients may use coumadin or heparin preparations
* have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation
* have a history of another primary malignancy ≤3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of the uterine cervix
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Oral contraceptives are not acceptable alone
* a contraindication to MRI
* are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to study treatment start
* unwilling or unable to comply with the protocol
* not affiliated to health system

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Radiographic response assessed by MRI analysis | after 1 year of treatment

SECONDARY OUTCOMES:
Radiographic response assessed by MRI analysis | At 2 years
Overall survival | At 2 years
Pain | At 2 years
Deficiency | At 2 years
Quality of life | At 2 years
adverse events | At 2 years
laboratory evaluations | At 2 years
measurement of vital signs | At 2 years
performance of physical examinations | At 2 years
all concomitant medications and therapies | At 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Wolkenstein, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Bissler JJ, McCormack FX, Young LR, Elwing JM, Chuck G, Leonard JM, Schmithorst VJ, Laor T, Brody AS, Bean J, Salisbury S, Franz DN. Sirolimus for angiomyolipoma in tuberous sclerosis complex or lymphangioleiomyomatosis. N Engl J Med. 2008 Jan 10;358(2):140-51. doi: 10.1056/NEJMoa063564. PMID 18184959
- [Derived] Zehou O, Ferkal S, Brugieres P, Barbarot S, Bastuji-Garin S, Combemale P, Valeyrie-Allanore L, Sbidian E, Wolkenstein P. Absence of Efficacy of Everolimus in Neurofibromatosis 1-Related Plexiform Neurofibromas: Results from a Phase 2a Trial. J Invest Dermatol. 2019 Mar;139(3):718-720. doi: 10.1016/j.jid.2018.09.016. Epub 2018 Oct 16. No abstract available. PMID 30339775